CLINICAL TRIAL: NCT06762327
Title: Ensartinib in the Treatment of ALK Positive or MET Exon 14 Skipping Anvanced Solid Tumors Excluded Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiaowei Wei, Associate chiefphysician, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV018
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ensartinib (Experimental)
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — ensartinib 225mg ,PO,QD,until disease progression or intolerable toxicity

SUMMARY:
In lung cancer, ensartinib is effective in improving the prognosis of ALK positive /MET exon 14 skipping patients. However, patients with ALK positive /MET14 exon skipping non-lung cancer solid tumors have limited treatment options in the absence of standard treatment. We hope to bring a new effective and safe treatment option to these patients more efficiently.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic solid tumors other than primary lung cancer
* Alk-positive or MET14 exon skipping mutation by IHC\FISH\NGS\RT-PCR
* Have no standard treatment after MDT discussion, or could not tolerate the standard treatment, or the patient refused the standard treatment
* Adequate liver and kidney function
* Adequate bone marrow function
* ECOG PS 0-3
* Female subjects should not be pregnant. All human subjects should able to comply with the required protocol and follow-up procedures, and able to receive oral medications Written informed consent provided

Exclusion Criteria:

* Active viral, bacterial, or fungal infection detected 2 weeks before enrollment
* Pregnancy or lactation
* receiving medications or herbal supplements with potent inducers of CYP3A4 (at least 3 weeks prior)
* Any severe or uncontrolled systemic illness, including uncontrolled Hypertension and active bleeding, any nonadherence that the investigator considered to be detrimental to study participation or adherence to the protocol, or active infections including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV)
* Ineligible cardiac function
* Interstitial lung disease, drug-induced interstitial lung disease, previous history of radiation pneumonitis requiring steroid therapy, or any evidence of active interstitial lung disease
* Lack of adequate bone marrow reserve or organ function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years
  time to progression or Intolerable toxicity occurred
Overall responce rate | 1year
  Proportion of patients with CR/PR response in the total population

SECONDARY OUTCOMES:
Disease control rate | 1year
  Proportion of patients with CR/PR/SD response in the total population
Overall survival | 3 years
  time to death
Duration of responce | 3 years
  time from first assessment of CR or PR to the first assessment of PD or death
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  The safety of Ensartinib treatment will be assessed according to CTCAE v5.0 criteria observed over the whole treatment period.